CLINICAL TRIAL: NCT01568060
Title: Assessment of Safety of GlaxoSmithKline (GSK) Biologicals' Combined Diphtheria-tetanus-acellular Pertussis-inactivated Poliovirus Vaccine, Infanrix-IPV When Administered According to the Approved Prescribing Information in Korea
Brief Title: Post-marketing Surveillance to Assess the Safety of Infanrix-IPV Vaccine Among Infants and Children in Korea
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114917
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Acellular Pertussis; Diphtheria; Tetanus; Poliomyelitis; Diphtheria-Tetanus-acellular Pertussis Vaccines
Keywords: Safety; Infanrix-IPV; Post-marketing surveillance; Diphtheria, tetanus, pertussis and poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis; Whooping Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Infanrix-IPV group: Infants and children who received at least one dose of Infanrix-IPV as a part of routine practice at a private clinic or hospital in korea
  Interventions: Other: Infanrix-IPV data collection

INTERVENTIONS:
Other: Infanrix-IPV data collection — Safety monitoring: recording of adverse events using diary cards and recording of serious adverse events using the latest version of Korea's Post-Marketing Surveillance Serious Adverse Event Reporting Form.

SUMMARY:
The purpose of this study is to collect safety information following routine vaccination with Infanrix-IPV among infants and children in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/legally acceptable representative(s) can and will comply with the requirements of the protocol.
* Korean male or female subjects who are eligible for the primary and/or booster doses of Infanrix-IPV according to the Korean Prescribing Information.
* Written or signed informed consent obtained from the parent(s)/ legally acceptable representative(s) of the child. Where parent(s)/ legally acceptable representatives are illiterate, the consent form will be countersigned by an impartial witness. Prior to enrollment of the subject into the post-marketing surveillance, the subject's parents/legally acceptable representatives will be requested to provide information regarding the enrollment of their child in a same/similar study previously. And prior to obtaining informed consent form, the investigator will check whether the subject is eligible for vaccination.

Exclusion Criteria:

* At the time of post-marketing surveillance (PMS) entry, the contraindications and precautions of use indicated in the local Prescribing Information should be checked and the subject must not be included in the PMS if there is any contraindication. Any changes in the locally approved Prescribing Information must be implemented immediately.
* Subjects who receive any investigational or non-licensed DTPa-IPV vaccine within 30 days prior to study start will not be enrolled.
* Child in care.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and children who receive at least one dose of Infanrix-IPV as a part of routine practice at a private clinic or hospital.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | During the 30-day (Day 0 - Day 29) follow-up period after each vaccine dose.
Occurrence of serious adverse events | Starting at Visit 1 in the post-marketing surveillance (PMS) up to 30 days (Day 0 to Day 29) after the last dose is administered in the PMS

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea

REFERENCES:
- [Background] Lee SM, Kim SJ, Chen J, Song R, Kim JH, Devadiga R, Kim YK. Post-marketing surveillance to assess the safety and tolerability of a combined diphtheria, tetanus, acellular pertussis and inactivated poliovirus vaccine (DTaP-IPV) in Korean children. Hum Vaccin Immunother. 2019;15(5):1145-1153. doi: 10.1080/21645515.2019.1572406. Epub 2019 Mar 19. PMID 30668217